CLINICAL TRIAL: NCT00623415
Title: Multicentric, Prospective, Double Blind, Randomized/Stratified, Placebo-controlled Pilot-study for Evaluation of Safety and Efficacy of Flupirtine add-on to Interferon-β1b on Neurodegeneration in Patients With Relapsing Remitting Multiple Sclerosis
Brief Title: Flupirtine as Oral Treatment in Multiple Sclerosis
Acronym: FLORIMS
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Bayer (Industry)
Responsible Party: Charite University, Berlin, Germany, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2006-005262-39
Record Dates: First submitted 2008-02-15; First posted 2008-02-26 (Estimated); Last update posted 2018-03-20 (Actual); Status verified 2017-12

CONDITIONS: Relapsing Remitting Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting | interventions — flupirtine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Verum (Active Comparator): flupirtine + interferon beta 1b
  Interventions: Drug: Flupirtine
- Placebo (Placebo Comparator): placebo + interferon beta 1b
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Flupirtine — 300 mg daily (divided in two doses)
  Arms: Verum
Drug: Placebo — twice daily
  Arms: Placebo

SUMMARY:
Flupirtine, a non-opioid analgesic drug, that has been shown to have additional neuroprotective functions, is given twice daily as an oral medication in patients with relapsing remitting multiple sclerosis over a period of 12 months. Neuroprotection is assessed by magnetic resonance imaging, magnetic resonance spectroscopy, optical coherence tomography, and clinical examination.

ELIGIBILITY:
Inclusion Criteria:

* Relapsing-remitting MS according to the revised McDonald-Criteria (2005)
* EDSS ≤ 4.0
* Stable treatment with Interferon-β1b for at least 6 months
* Sufficient birth control (Pearl-Index <1)

Exclusion Criteria:

* Any other MS-course than RRMS
* Clinically relevant gastrointestinal disease
* Clinically relevant pulmonary, cardiological, infectious or CNS-disease
* Clinically relevant disease of liver or bile system, pathological value for transaminases, gamma-GT or bilirubin.
* Hepatitis (except uncomplicated hepatitis A with complete remission
* Clinically relevant dysfunction of kidneys (creatinine >180 µmol/l) or bone marrow (HB < 8.5 g/dl, WBC < 2.5/nl thrombocytes < 125/nl)
* Myasthenia gravis
* Oral anticoagulation (phenprocoumon)
* Treatment with carbamazepine or paracetamol
* Drug or alcohol abuse
* Pregnancy or lactation period
* Treatment at any time before or during study with complete lymphoradiation, monoclonal antibodies (e.g. anti-CD4, Campath 1H, natalizumab), mitoxantrone, cyclophosphamide, cyclosporin, azathioprine
* Treatment within 6 months before randomization with any other immunomodulatory substance than interferon-β1b or intravenous methylprednisolone

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2007-12; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Cumulative number of new T2-hypertensive lesions on cranial magnetic resonance imaging (MRI) | 12 months

SECONDARY OUTCOMES:
Cerebral atrophy (brain parenchymal fraction) | 12 months
Number of new and total gadolinium(Gd)-enhancing lesions | 12 months
Disease progression (measured by Expanded Disability Status (EDSS), Multiple Sclerosis Functional Composite (MSFC)) | 12 months
Retinal nerve fiber layer thickness, assessed by Optical coherence tomography | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Friedemann Paul, MD, Principal Investigator — NeuroCure Clinical Research Center, Charité Berlin, Germany
Locations (4):
- Germany (4):
  - NeuroCure Clinical Research Center, Charité Berlin, Berlin
  - Carl-Thiem-Clinic Cottbus, Cottbus
  - University of Göttingen, Department of Neurology, Göttingen
  - University of Ulm, Department of Neurology, Ulm